CLINICAL TRIAL: NCT01846884
Title: Urine Sample Processing Study:Analysis of Fresh Versus Frozen Urine Samples From Critically Ill Subjects
Brief Title: Specimen Stability Study
Status: Completed | Type: Observational
Sponsor: Astute Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Opal
Record Dates: First submitted 2013-04-29; First posted 2013-05-06 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To collect and process urine samples from critically ill subjects for use in assessing the effects of various urine sample freezing and storage conditions on biomarker test results.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 21 years of age or older
2. Subjects must be enrolled (first study-specific sample collection) within 24 hours of ICU admission

   * Subjects enrolled from ED or Floor must be admitted to the ICU within 24 hours of enrollment
   * Subjects enrolled in the ICU must have been admitted to the ICU or transferred into the study ICU from another ICU no more than 24 hours prior to enrollment
3. Expected to remain in the ICU for at least 48 hours after enrollment
4. Use of indwelling urinary catheter as standard care expected for at least 48 hours after enrollment
5. Subject (or authorized representative)able and willing to provide written informed consent for study participation

Exclusion Criteria:

1. Special populations including children, pregnant women, and prisoners
2. Previous renal transplantation
3. Already receiving dialysis (either acute or chronic) or in imminent need of dialysis at the time of enrollment
4. Known infection with human immunodeficiency virus (HIV) or active hepatitis (acute or chronic)
5. Subjects with a history of chronic kidney disease (CKD) without a baseline serum creatinine value (baseline within 6 months of enrollment)
6. Previously provided a urine sample and enrolled in this study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically-ill adult subjects at risk for acute kidney injury.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Specimen handling and stability, for example, effect of temperature on biomarker results. There are no primary clinical outcomes. | 6 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - La Mesa, California
  - Honolulu, Hawaii
  - Idaho Falls, Idaho
  - Las Vegas, Nevada
  - Port Jefferson, New York
  - Greenville, North Carolina

REFERENCES:
- [Derived] Hoste EA, McCullough PA, Kashani K, Chawla LS, Joannidis M, Shaw AD, Feldkamp T, Uettwiller-Geiger DL, McCarthy P, Shi J, Walker MG, Kellum JA; Sapphire Investigators. Derivation and validation of cutoffs for clinical use of cell cycle arrest biomarkers. Nephrol Dial Transplant. 2014 Nov;29(11):2054-61. doi: 10.1093/ndt/gfu292. Epub 2014 Sep 18. PMID 25237065